CLINICAL TRIAL: NCT02883205
Title: Diagnosis of Fabry Disease: Impact of an Educational Brochure Intended for Cardiologist
Acronym: TARIFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-060
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The cardiac Fabry disease are early, frequent and severe, dominated by the frequency of left ventricular hypertrophy. They are responsible for a high morbidity and mortality, reducing life expectancy of 15 to 20 years for men. Fabry disease and heart attacks are still diagnosed late. This delay in diagnosis is due to the non-specificity of clinical, electrocardiographic and echocardiographic disease, but also by a certain ignorance of this pathology in the medical community. The importance of early diagnosis of Fabry disease and heart disease is well established: enzyme replacement therapy is most effective when instituted early, before the onset of irreversible damage such as fibrosis. With the blotter, we now have a simple and robust screening tool for Fabry disease, achievable consultation. Targeted educational interventions to physicians have shown their effectiveness in improving the screening and diagnosis of rare diseases. We offer a prospective observational type before / after study, which aims to assess the value of an educational brochure for cardiologists to improve the screening and diagnosis of Fabry disease in Normandy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with left ventricular hypertrophy of unknown etiology or of sarcomeric MHC pace, followed in Normandy, has given its consent to the search of Fabry disease

Criteria Exclusion:

* Patients under 18 years patient refusal to participate in the study. Lack of consent to the search of Fabry disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with left ventricular hypertrophy of unknown etiology or of sarcomeric MHC pace, followed in Normandy, has given its consent to the search of Fabry disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of new cases of Fabry disease diagnosed a year after distribution of educational brochure cardiologists | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Labombarda, MD, Principal Investigator — Caen HU
Locations (1):
- Fabien, Caen, France

IPD SHARING:
Plan to Share IPD: No